CLINICAL TRIAL: NCT02128984
Title: Clinical Study With an Enteral Formula With Symbiotic and DHA for Malnourished Children
Acronym: VITJUNIOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratorios Ordesa (Industry)
Collaborators: Quantum Experimental (Unknown); Peruvian Clinical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VIT-2572-011
Record Dates: First submitted 2014-03-28; First posted 2014-05-01 (Estimated); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Cystic Fibrosis; Failure to Thrive; Malnutrition
Keywords: Malnutrition; Dietary supplement; Nutritional supplement; Symbiotic formula; DHA; Cystic Fibrosis; Failure to Thrive
MeSH Terms: conditions — Cystic Fibrosis; Failure to Thrive; Malnutrition | interventions — Antioxidants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitafos Junior (Experimental): Symbiotic Formula with DHA and antioxidants
  Interventions: Dietary Supplement: Symbiotic Formula with DHA and antioxidants
- Standard Formula (Active Comparator): Standard isocaloric and isonitrogenous formula.
  Interventions: Dietary Supplement: Standard Formula

INTERVENTIONS:
Dietary Supplement: Symbiotic Formula with DHA and antioxidants — 6 months intervention.
  Other Names: Vitafos Junior
  Arms: Vitafos Junior
Dietary Supplement: Standard Formula — 6 months intervention.
  Arms: Standard Formula

SUMMARY:
The purpose of this study is to determine whether a nutritional supplement is effective in the treatment of malnutrition in pediatric patients with failure to thrive or cystic fibrosis.

DETAILED DESCRIPTION:
This is a multicenter, controlled, randomized, prospective, parallel-group, double-blind study to evaluate the effect of a nutritional supplement on nutritional status in children with failure to thrive or cystic fibrosis. Patients will be randomized to receive either a symbiotic formula with DHA and antioxidants or a standard formula.

ELIGIBILITY:
Inclusion Criteria:

* Malnutrition (P / T <-1 SD) by intake deficit without organic disease (failure to thrive) and / or patients diagnosed with Cystic Fibrosis).
* Age >= 1 year.
* Stable patients
* No antibiotherapy in the last 30 days
* Inform consent signed (parent/legal representative)

Exclusion Criteria:

* Patients with allergy / intolerance to cow's milk proteins
* Metabolically unstable patient
* Patients with metabolic intolerance to carbohydrates
* Patients with severe disease in the last 30 days

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2012-01; Primary Completion 2015-02 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Changes in inflammatory response | At 3rd and 6th months
  Differences in faecal calprotectin's levels after 3rd and 6th months of treatment.

SECONDARY OUTCOMES:
Changes in nutritional status | At 3rd and 6th months
  Differences measured by changes in weight, height, growth Z-scores, fat body mass and lean body mass.
Changes in microbiota profile | At 3rd and 6th months
  Differences measured by changes in faecal microbiota composition.
Changes in Interleukin levels | At 6th month
  Differences in faecal interleukin levels. Only for cystic fibrosis patients.
Incidence of Infections | At 1st, 3rd and 6th months
  Episodes of infections during the study period

OTHER OUTCOMES:
Tolerability of the formula | At 1st, 3rd and 6th months
  Tolerability to the formula in both groups

CONTACTS AND LOCATIONS:
Locations (8):
- Instituto Nacional de Salud del Niño, Lima, Breña, Peru
- Spain (7):
  - Hospital de Henares, Coslada, Madrid
  - Hospital Universitario Santa Lucía, Cartagena, Murcia
  - Hospital de Torrecárdenas, Almería
  - Hospital Puerta del Mar, Cadiz
  - Hospital Universitario La Paz, Madrid
  - Hospital Virgen Macarena, Seville
  - Hospital Universitario Miguel Servet, Zaragoza